CLINICAL TRIAL: NCT04273958
Title: Impact of the Use of Virtual Reality on Pain and Anxiety Caused by Invasive Medical Procedures in the Emergency Department
Brief Title: Virtual Reality During Invasive Medical Procedures in an Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olivier Hugli (Other)
Collaborators: University of Lausanne (Other)
Responsible Party: Sponsor-Investigator, Olivier Hugli, Professor, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019-02276
Record Dates: First submitted 2020-02-12; First posted 2020-02-18 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Pain; Anxiety; Virtual Reality
Keywords: pain; virtual reality; anxiety; emergency department; procedural pain
MeSH Terms: conditions — Pain; Anxiety Disorders; Emergencies; Pain, Procedural

STUDY DESIGN:
Intervention Model Description: Each patient will be randomized in a 1:1 ratio between the two arms of the study
Who Masked: Investigator
Masking Description: The study will be a randomized controlled study. In order to minimize bias, one investigator will randomize the patient to one of the two groups, set up the medium to which the patient is assigned, and be present during the procedure. Patients will evaluate their pain and anxiety levels themselves using an electronic tablet, without the help of the investigator.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality (Experimental): The intervention will consist of the use of a virtual reality helmet during the painful medical procedure. The content has been developed by a private company with the goal of providing a relaxing and soothing exploration of a virtual world.
  Interventions: Device: Virtual reality helmet
- Computer screen (Active Comparator): The comparator will consist in the screening of the same virtual world on the computer screen.
  Interventions: Device: Computer screen

INTERVENTIONS:
Device: Virtual reality helmet — During a painful procedure, the patient will watch a virtual world in a virtual reality helmet, while wearing a noise-canceling headset with soothing music.
  Arms: Virtual reality
Device: Computer screen — During a painful procedure, the patient will watch the same virtual world, while wearing a noise-canceling headset with the same soothing music.
  Arms: Computer screen

SUMMARY:
This randomized controlled study aims to investigate whether, during a painful medical procedure in an emergency department (ED), the diffusion of a virtual environment through a virtual reality (VR) headset worn by the patient has a greater impact on the patient's pain and anxiety levels than the diffusion of an identical environment through a computer screen. The study design allows differentiating the impact of the medium from that of the media. The feeling of telepresence of patients in both groups and its association with the impact of the medium will also be investigated.

In addition, this study aims to explore whether the wearing of VR headphones is considered comfortable and acceptable by patients.

DETAILED DESCRIPTION:
Consultation in a hospital ED and the provided treatments are stressful, as it usually results from an unexpected event that has a negative impact on health. Also, an ED is a noisy and chaotic environment, which can increase anxiety and pain sensitivity related to certain medical procedures. Indeed, the conditions under which medical and surgical procedures are performed have an impact on the patient's experience: pain can be more intense if the patient is stressed and focused on the medical procedure. The well-being of patients, especially during these invasive medical procedures, can be improved by adjusting the conditions in which the procedure is performed.

The literature and clinical observations show that distraction is a very effective non-pharmacological strategy to reduce pain and anxiety. The use of measures such as television, music or other audiovisual media has been shown to decrease pain during painful medical procedures in ED. The perception of pain competes with other stimuli, whether sensory or psychological. This competition is all the more effective as the number of senses involved and their intensity increases. However, these traditional media have little distractive power. They capture partially the patient's attention and the patient can easily refocus on the ongoing medical procedure.

These traditional media do not produce an immersive experience. According to this principle, the analgesic effect of VR is expected to be greater than that provided by passive distractions such as watching a film on television, as demonstrated during wound dressing replacement in burned patients. Also, the patient's emotional state plays a role in her/his distractibility during a procedure. Therefore, the ideal distractive method should involve a maximum of senses (vision/hear/touch/...) and affects the patient's emotions to compete with the unpleasant stimulus.

VR is a recent technology that offers a multi-sensory (vision, hearing), immersive and three-dimensional experience. It offers an active immersion in a virtual world, letting the patient navigate in a virtual world, leading to a greater perceived presence in this virtual environment (telepresence). Telepresence allows the patient to be a co-constructor of the experience. It differentiates VR from other cognitive and distractive techniques. VR can thus distract patients more effectively from the conditions under which they receive their treatment by procuring a superior distraction. However, studies on the impact of VR during invasive or painful procedures have left some unanswered questions that limit its unrestricted use in the ED :

* Most of the studies have been conducted in children.
* Different technologies have been used by different studies, precluding direct comparisons between studies;
* There are few data on the impact of VR applied in an emergency department with adult patients;
* The differentiation between the effect of the media (images used) and the effect of the medium (technology used) is often neglected; In this study, the investigators will attempt to demonstrate the potential superiority of VR, using a commercial VR device projecting a virtual environment designed specifically for medical use by a private company, and available to any group or ED wishing to apply this technology. The investigators will include adult patients requiring a painful medical procedure. In addition, patients will be randomized between two groups, both exposed to the same virtual environment (media) but screened in two different technologies (medium).

ELIGIBILITY:
Inclusion Criteria:

* Patient whose care requires a medical procedure (suture, cast placement and repositioning, fracture reduction, paracentesis, thoracocentesis and lumbar puncture).

Exclusion Criteria:

* Unstable patient (e.g., admitted to the intensive care unit or deemed unstable by the physician in charge);
* Patients without decision-making capacity or with whom it is difficult to communicate:
* Altered mental status (e.g., cognitive impairment, mental retardation, acute confusional state, acute psychosis).
* Intoxication,
* Drug abuse
* Patient unable to communicate in French at a level sufficient to give informed consent and answer questions about pain and anxiety;
* Patient who is hard of hearing;
* Patient unable to see films on screen or in VR due to vision problems (e.g., blindness or without his/her glasses).
* Patients unable to understand the use of the EVA strips;
* Part of the body where the altered procedure is to be performed (e.g. sensitivity disorder, lymphedema...)
* Patient with a head injury that prevents the use of RV helmet;
* Intended use of sedation analgesia with a dissociative agent (midazolam, ketamine, propofol).
* Incarcerated patient;
* Patient transferred from another hospital;
* Patient who participated in this study at a previous consultation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Pain reduction | Pain intensity will be assessed immediately before and immediately after the procedure.
  The primary outcome of this study will be the patients' self-assessment of their pain intensity by Visual Analog Scale (VAS) on a 100-mm ruler during the procedure in the emergency department. The ruler will be presented to the patients on a digital tablet, and the patients will place the slider along the 100-mm line anchored at each end by the two labels "no pain" / "worst pain imaginable". The numerical value measured in millimeters will be automatically integrated into the electronic Case Report Form (CRF).
Anxiety reduction | Anxiety intensity will be assessed immediately before and immediately after the procedure.
  The primary outcome of this study will be the patients' self-assessment of their anxiety intensity by Visual Analog Scale (VAS) on a 100-mm ruler during the procedure in the emergency department. The ruler will be presented to the patients on a digital tablet, and the patients will place the slider along the 100-mm line anchored at each end by the two labels "no anxiety" / "worst anxiety imaginable". The numerical value measured in millimeters will be automatically integrated into the electronic Case Report Form (CRF).

SECONDARY OUTCOMES:
Telepresence | Telepresence feeling will be assessed immediately at the end of the procedure.
  The first secondary outcome of this study will be patients' assessment of their telepresence perception using the iGroup Presence Questionnaire.
Level of dissociation | Dissociation will be assessed immediately at the end of the procedure.
  The next secondary outcomes will be patients' assessment of their level of dissociation by a specific question; it will also be measured by testing the understanding of the procedure by a Visual Analog Scale (VAS) on a 100-mm ruler. The ruler will be presented to the patients on a digital tablet, and the patients will place the slider along the 100-mm line. The ruler for the understanding of the procedure will be anchored by the terms "no understanding" / "complete understanding".The numerical value measured in millimeters will be automatically integrated into the electronic Case Report Form (CRF).
Patient's acceptance of the technology | Acceptance will be assessed immediately at the end of the procedure.
  Patients'acceptance will be measured by a Visual Analog Scale (VAS) on a 100-mm ruler. The ruler will be presented to the patients on a digital tablet, and the patients will place the slider along the 100-mm line. The ruler for the acceptance of the technology will be anchored by the terms "not acceptable" / "completely acceptable".The numerical value measured in millimeters will be automatically integrated into the electronic Case Report Form (CRF).
Patient's comfort with the technology | Comfort will be assessed immediately at the end of the procedure.
  Patient's comfort with the technology will be measured by a Visual Analog Scale (VAS) on a 100-mm ruler. The ruler will be presented to the patients on a digital tablet, and the patients will place the slider along the 100-mm line. The ruler for the comfort with the technology will be anchored by the terms "very comfortable" / "very uncomfortable".The numerical value measured in millimeters will be automatically integrated into the electronic Case Report Form (CRF).
Motion sickness | Motion sickness will be assessed immediately at the end of the procedure.
  Motion sickness is one of the side-effect of a virtual reality headset. Patient's motion sickness will be measured by a Visual Analog Scale (VAS) on a 100-mm ruler. The ruler will be presented to the patients on a digital tablet, and the patients will place the slider along the 100-mm line. The ruler for the comfort with the technology will be anchored by the terms "no motion sickness" / gratest motion sickness imaginable".The numerical value measured in millimeters will be automatically integrated into the electronic Case Report Form (CRF).
Perception by physicians of this technology | Perception by physicians of this technology will be assessed immediately at the end of the procedure.
  Physicians' perception of the usefulness provided by the technology will be assessed by two questions. The first question will address the help provided by the technology (Did the technology used help you during the procedure? Possible answers will be yes, no, neutral). The second question will enquire if the question has hindered the physician (Did the technology used hinder you during the procedure?Possible answers will be yes, no, neutral).

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Hugli, MD, MPH, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bantick SJ, Wise RG, Ploghaus A, Clare S, Smith SM, Tracey I. Imaging how attention modulates pain in humans using functional MRI. Brain. 2002 Feb;125(Pt 2):310-9. doi: 10.1093/brain/awf022. PMID 11844731
- [Background] Downey LV, Zun LS. The impact of watching cartoons for distraction during painful procedures in the emergency department. Pediatr Emerg Care. 2012 Oct;28(10):1033-5. doi: 10.1097/PEC.0b013e31826cac1a. PMID 23023471
- [Background] Sikka N, Shu L, Ritchie B, Amdur RL, Pourmand A. Virtual Reality-Assisted Pain, Anxiety, and Anger Management in the Emergency Department. Telemed J E Health. 2019 Dec;25(12):1207-1215. doi: 10.1089/tmj.2018.0273. Epub 2019 Feb 20. PMID 30785860
- [Background] Jeffs D, Dorman D, Brown S, Files A, Graves T, Kirk E, Meredith-Neve S, Sanders J, White B, Swearingen CJ. Effect of virtual reality on adolescent pain during burn wound care. J Burn Care Res. 2014 Sep-Oct;35(5):395-408. doi: 10.1097/BCR.0000000000000019. PMID 24823326
- [Background] Toledo Del Castillo B, Perez Torres JA, Morente Sanchez L, Escobar Castellanos M, Escobar Fernandez L, Gonzalez Sanchez MI, Rodriguez Fernandez R. [Reducing the pain in invasive procedures during paediatric hospital admissions: Fiction, reality or virtual reality?]. An Pediatr (Engl Ed). 2019 Aug;91(2):80-87. doi: 10.1016/j.anpedi.2018.10.019. Epub 2019 Jan 21. Spanish. PMID 30679136
- [Background] Garrett B, Taverner T, Gromala D, Tao G, Cordingley E, Sun C. Virtual Reality Clinical Research: Promises and Challenges. JMIR Serious Games. 2018 Oct 17;6(4):e10839. doi: 10.2196/10839. PMID 30333096
- [Background] Vanhaudenhuyse A, Ledoux D, Gosseries O, Demertzi A, Laureys S, Faymonville ME. CAN SUBJECTIVE RATINGS OF ABSORPTION, DISSOCIATION, AND TIME PERCEPTION DURING "NEUTRAL HYPNOSIS" PREDICT HYPNOTIZABILITY?: An exploratory study. Int J Clin Exp Hypn. 2019 Jan-Mar;67(1):28-38. doi: 10.1080/00207144.2019.1553765. PMID 30702397
- [Background] Li SF, Greenwald PW, Gennis P, Bijur PE, Gallagher EJ. Effect of age on acute pain perception of a standardized stimulus in the emergency department. Ann Emerg Med. 2001 Dec;38(6):644-7. doi: 10.1067/mem.2001.119849. PMID 11719743
- [Background] Singer AJ, Richman PB, Kowalska A, Thode HC Jr. Comparison of patient and practitioner assessments of pain from commonly performed emergency department procedures. Ann Emerg Med. 1999 Jun;33(6):652-8. PMID 10339680
- [Background] Lang EV, Tan G, Amihai I, Jensen MP. Analyzing acute procedural pain in clinical trials. Pain. 2014 Jul;155(7):1365-1373. doi: 10.1016/j.pain.2014.04.013. Epub 2014 Apr 13. PMID 24731852
- [Background] Page MG, Katz J, Stinson J, Isaac L, Martin-Pichora AL, Campbell F. Validation of the numerical rating scale for pain intensity and unpleasantness in pediatric acute postoperative pain: sensitivity to change over time. J Pain. 2012 Apr;13(4):359-69. doi: 10.1016/j.jpain.2011.12.010. Epub 2012 Mar 15. PMID 22424915
- [Derived] Bosso L, Espejo T, Taffe P, Caillet-Bois D, Christen T, Berna C, Hugli O. Analgesic and Anxiolytic Effects of Virtual Reality During Minor Procedures in an Emergency Department: A Randomized Controlled Study. Ann Emerg Med. 2023 Jan;81(1):84-94. doi: 10.1016/j.annemergmed.2022.04.015. Epub 2022 May 28. PMID 35641354